CLINICAL TRIAL: NCT00175396
Title: A Randomized Phase III Study Comparing Androgen Suppression and Elective Pelvic Nodal Irradiation Followed by High Dose 3-D Conformal Boost Versus Androgen Suppression and Elective Pelvic Nodal Irradiation Followed by 125-Iodine Brachytherapy Implant Boost for Patients With Intermediate and High Risk Localized Prostate Cancer
Brief Title: Androgen Suppression Combined With Elective Nodal and Dose Escalated Radiation Therapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H04-60050; H04-60050
Record Dates: First submitted 2005-09-11; First posted 2005-09-15 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Prostate Cancer
Keywords: ASCENDE-RT
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy; nilutamide; bicalutamide; Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Procedure: Androgen suppression, radiotherapy
- 2 (Experimental)
  Interventions: Procedure: Androgen suppression, radiotherapy, iodine 125 brachytherapy

INTERVENTIONS:
Procedure: Androgen suppression, radiotherapy — Total of 12 months of androgen suppression. 8 months after the start of androgen suppression 4.2-5 weeks external beam radiation (46 Gy in 23 equal fractions) followed by an external beam radiation boost lasting 3.2-4 weeks (32 Gy in 16 equal fractions).
  Other Names: Androgen suppression: non-steroidal androgen (any of flutamide, nilutamide or bicalutamide (bicalutamide is almost always used).; LHRH monotherapy: buserelin acetate or leuprolide acetate.
  Arms: 1
Procedure: Androgen suppression, radiotherapy, iodine 125 brachytherapy — Total of 12 months of androgen suppression. 8 months after the start of androgen suppression 4.2-5 weeks external beam radiation (46 Gy in 23 equal fractions) followed by iodine 125 brachytherapy carried out 14-25 days after the last external beam treatment.
  Arms: 2

SUMMARY:
The purpose of this trial is to compare two similar treatments for patients diagnosed with prostate cancer. The two treatment arms being compared are: (Standard Arm) hormone therapy, which will prevent the production of the male hormone, testosterone, by the testicles, and pelvic external beam radiation therapy (EBRT) followed by a high-dose, conformal EBRT boost versus (Investigational Arm) hormone therapy and pelvic EBRT followed by a brachytherapy boost (implantation of radioactive iodine sources or "seeds" into the prostate).

The hypothesis of this trial is that more patients may experience 5 year actuarial freedom from biochemical recurrence of their prostate cancer following treatment with the investigational arm. Biochemical failure is declared on the date when the post treatment prostate specific antigen (PSA) is > 2 ng/mL above the lowest level previously recorded.

DETAILED DESCRIPTION:
Patients will be randomly assigned with equal probability to one or two treatment arms, Arm 1 or Arm 2, where the interventions associated with these Arms are as follows:

Arm 1:

Neoadjuvant, concurrent and adjuvant androgen suppression, elective pelvic nodal irradiation (EPNI), high dose conformal EBRT boost to the prostate, and appropriate secondary interventions at failure.

Arm 2:

Neoadjuvant, concurrent and adjuvant androgen suppression, elective pelvic nodal irradiation (EPNI), permanent 125-Iodine brachytherapy boost to the prostate, and appropriate secondary interventions at failure.

If a patient is assigned to Arm 1, the radiation oncologist will initiate androgen suppression and monitor clinical and biochemical response. After an 8-month duration of neoadjuvant androgen suppression, the patient will undergo a course of elective pelvic nodal irradiation (EPNI) to a volume encompassing the prostate gland, seminal vesicles and regional lymph nodes. The pelvic irradiation will be followed by a dose-escalated 3-D conformal EBRT boost to the prostate with appropriate margins. The total radiation dose to the regional lymphatics is 46 Gy and prostate dose is 78 Gy at the ICRU reference point with a minimum dose to the PTV of > 74 Gy. Androgen suppression is maintained throughout radiation therapy and following the completion of radiation therapy until the patient has received a total duration of androgen suppression of 12 months including the neoadjuvant phase.

If the patient is assigned to Arm 2, the radiation oncologist will initiate androgen suppression and monitor clinical and biochemical response. After an 8-month duration of neoadjuvant androgen suppression, the patient will undergo a course of elective pelvic nodal irradiation (EPNI) to a volume encompassing the prostate gland, seminal vesicles and regional lymph nodes. The total radiation dose to the regional lymphatics is 46 Gy. Two weeks following the completion of the pelvic irradiation, the patient will undergo a permanent 125-Iodine brachytherapy prostate implant at the facilities of the participating institution by a team of healthcare professionals lead by a Radiation Oncologist with experience in prostate brachytherapy. To be eligible to participate, the institution must have done at least 25 cases of prostate brachytherapy with stranded sources. The minimal peripheral dose (MPD) to the prostate gland from the implant will be 115 Gy. A modified peripheral loading technique will be used in an effort to maintain the periurethral dose to < 150% of the MPD. Androgen suppression is maintained throughout radiation therapy until the patient has received a total duration of androgen suppression of 12 months including the neoadjuvant phase.

All patients randomized are part of the analysis. The patient remains on study whether or not protocol treatment defined for the assigned arm is completed. The end of the primary intervention is defined as 18 months following the start of neoadjuvant androgen suppression in both arms.

Secondary Objectives:

Overall survival, metastasis-free survival, pathological local control, incidence of acute and late side effects and complications associated with the treatment interventions, effect of the planned interventions on QOL and rate of testosterone recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically-proven prostate cancer stage T1c -T3a (UICC 1997).
2. Patients with clinically organ-confined disease must meet the Canadian consensus definition of intermediate risk disease (i.e any one or more of: CS = T2b [UICC1997 = bilateral palpable intra-capsular disease], GS = 7, or iPSA >10 and 20).
3. Patients with Gleason sum 8 and/or PSA > 20 must have a CT pelvis, and nuclear medicine bone scan showing no evidence of nodal (N0) or distant metastases (M0).
4. Registration must occur within 36 weeks of biopsy.
5. Patients with clinical or pathological evidence of seminal vesicle invasion (stage T3b) or involvement of adjacent pelvic organs/structures (stage T4) are not eligible.
6. Pre-intervention PSA must not exceed 40 ng ml-1.
7. Patients must have a chest x-ray and the following blood tests within four weeks of registration: PSA, PAP, testosterone, CBC, electrolytes, BUN, creatinine, AST, LDH and alkaline phosphatase. Patients with values for one or more of these tests that fall outside the normal range will not necessarily be ineligible, however, their eligibility will need to be reviewed by the study coordinator.
8. Patients must have an ECG within four weeks of registration. Patients with ECGs judged to be significantly abnormal require a consultation with a cardiologist to ascertain their suitability for general or spinal anesthesia.
9. Patients judged clinically to have a prostate volume > 65 cm3 prior to starting androgen suppression must have a transrectal ultrasound for volume estimation. Patients with TRUS prostate volumes > 75 cm3 prior to starting androgen suppression are not eligible for the study.
10. Patients may have been started on neoadjuvant androgen suppression prior to registration provided:

    * there is documentation of pre-treatment PSA and
    * in the case of patients with iPSA >20 and/or Gleason sum 8, a bone scan and CT pelvis were done prior to or within 4 weeks after starting neoadjuvant androgen suppression.
11. Patients must not have received prior surgical treatment for prostate cancer including transurethral resection of the prostate (TURP), transurethral resection of the bladder neck (TURB), cryotherapy, laser ablation, or microwave therapy.
12. Patients should have an estimated life expectancy of at least 5 years with an ECOG performance status of 0-2.
13. Patients may not have received prior radiation therapy to the pelvis.
14. Patients must be fit for general or spinal anesthetic.
15. Patients on Coumadin therapy must be able to stop the therapy safely for at least 12 days. Documentation as to the safety of such an interruption in anticoagulation therapy must be provided by an appropriate specialist physician (usually a cardiologist or hematologist).
16. Patients must be judged to have no contraindication to high dose pelvic irradiation or LHRH agonist therapy.
17. Cancer survivors are eligible providing that all three of the following criteria are met:

    * The patient has undergone potentially curative therapy for all prior malignancies.
    * There has been no evidence of recurrence for at least five years following potentially curative therapy. (For non-melanoma skin cancer the five-year requirement does not apply.)
    * The patient is considered by the treating physician to be at low risk of recurrence from prior malignancies.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2004-05; Primary Completion 2011-12 (Actual); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
The primary end point of this trial is 5 year actuarial freedom from biochemical recurrence (5 year bNED) using the Houston definition of biochemical failure. | 5 years

SECONDARY OUTCOMES:
This trial is also intended to determine overall survival, metastasis-free survival, pathological local control, incidence of acute and late side effects and complications associated with the treatment interventions, effect of the planned interventions. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: William J Morris, MD, Principal Investigator — University of British Columbia
Locations (1):
- BC Cancer Agency, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Morris WJ, Pickles T, Keyes M. Using a surgical prostate-specific antigen threshold of >0.2 ng/mL to define biochemical failure for intermediate- and high-risk prostate cancer patients treated with definitive radiation therapy in the ASCENDE-RT randomized control trial. Brachytherapy. 2018 Nov-Dec;17(6):837-844. doi: 10.1016/j.brachy.2018.08.008. Epub 2018 Sep 21. PMID 30245169
- [Derived] Rodda S, Morris WJ, Hamm J, Duncan G. ASCENDE-RT: An Analysis of Health-Related Quality of Life for a Randomized Trial Comparing Low-Dose-Rate Brachytherapy Boost With Dose-Escalated External Beam Boost for High- and Intermediate-Risk Prostate Cancer. Int J Radiat Oncol Biol Phys. 2017 Jul 1;98(3):581-589. doi: 10.1016/j.ijrobp.2017.02.027. Epub 2017 Feb 21. PMID 28581398
- [Derived] Rodda S, Tyldesley S, Morris WJ, Keyes M, Halperin R, Pai H, McKenzie M, Duncan G, Morton G, Hamm J, Murray N. ASCENDE-RT: An Analysis of Treatment-Related Morbidity for a Randomized Trial Comparing a Low-Dose-Rate Brachytherapy Boost with a Dose-Escalated External Beam Boost for High- and Intermediate-Risk Prostate Cancer. Int J Radiat Oncol Biol Phys. 2017 Jun 1;98(2):286-295. doi: 10.1016/j.ijrobp.2017.01.008. Epub 2017 Jan 6. PMID 28433432